CLINICAL TRIAL: NCT02665091
Title: Impact of Peer Education Program on HIV/AIDS Related Sexual Behaviors of Secondary School Students in Rural Communities, India: a Quasi-experimental Study.
Brief Title: Peer Education Program for HIV/AIDS Related Sexual Behaviors of Secondary School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: nmp/22189
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peer Education Group (Experimental): Group was self compared after the intervention
  Interventions: Behavioral: Peer Education Program

INTERVENTIONS:
Behavioral: Peer Education Program

SUMMARY:
Worldwide, about 50% of all new cases of HIV occur in youth between age 15 and 24 years. Studies in various countries show that both out of school and in school adolescents and youth are engaged in risky sexual behaviors. Peer-based interventions have become a common method to effect important health-related behavior changes and address the HIV/AIDS pandemic. This study therefore aimed to evaluate the effectiveness of peer education in improving HIV knowledge, attitude, and preventive practices among in-school adolescents

ELIGIBILITY:
Inclusion Criteria:

* at least 14 years of age;
* non-injecting use of heroin, cocaine or crack cocaine in the last six months;
* test HIV antibody negative;
* agree to provide specimens for testing (HIV, HBV and pregnancy) and be willing to learn the results of these tests;
* willing to return for visits at 1, 6, and 9 months post-enrollment;
* willing and able to provide informed consent.

Exclusion Criteria:

* history of injection drug use in the previous 3 years;
* pregnant;

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 560 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Knowledge score of HIV | From baseline to 6 Months

SECONDARY OUTCOMES:
willingness to HIV testing | From Baseline to 6 Months
willingness to participate in HIV counseling services | From Baseline to 6 Months
frequency of use of Condoms | From baseline to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hitesh Nayak, Principal Investigator — NMP Medical Research Institute; Neha Sharma, PhD, Study Director — Warwick Research Services; Valerie Murray, MA, Study Chair — Goldington Family Centre, UK

IPD SHARING:
Plan to Share IPD: Yes
YES